CLINICAL TRIAL: NCT02511964
Title: Effect of Six Running Sessions of High Intensity Interval Training in Different Slopes on Aerobic Performance: a Randomized Controlled Trial
Brief Title: High Intensity Interval Training in 1% or 10% Slope
Acronym: Slope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGF 01
Record Dates: First submitted 2015-07-11; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Aerobic Exercise; HIT,; VO2Max; Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interval Training at 1% incline (Experimental): Six Sessions of High Intensity Interval Running (100% VO2Max) at 1% incline; Group metabolically balanced.
  Interventions: Behavioral: Interval Training at 1% Incline
- Interval Training at 10% incline (Experimental): Six Sessions of High Intensity Interval Running (100% VO2Max) at 10% incline; Group metabolically balanced.
  Interventions: Behavioral: Interval Training at 10% Incline
- Control (No Intervention): Only Dependent Variables Measures

INTERVENTIONS:
Behavioral: Interval Training at 1% Incline — Six Sessions of Running at 1% incline
  Other Names: HIT in 1% Slope; HIIT in 1% Slope
  Arms: Interval Training at 1% incline
Behavioral: Interval Training at 10% Incline — Six Sessions of Running at 10% incline
  Other Names: HIT in 10% Slope; HIIT in 10% Slope
  Arms: Interval Training at 10% incline

SUMMARY:
The objective was to determine the effect of six running sessions of high intensity interval training (HIIT) at 1% and 10% incline on VO2max, peak of velocity (VPeak), and time limit of 1% (TLim1%) and 10% (TLim10%) of inclination, as well as the influence of the specificity of training on performance in the different inclines.

DETAILED DESCRIPTION:
Our study is assuming greater activation / muscle overload coming from the uphill running. Accordingly, we believe that in a parallel-group design (1% or 10% gradient) established in controlled and randomized way we could answer the hypothesis that muscle overload provide superior gains to VO2max and aerobic performance. Moreover, considering the first hyphotesis, such developments on the running at 10% slope also promote significant gains in climb performance and also in the plan. Unlike the speculate that the gains from the 1% training does not help performance a 10% incline.

ELIGIBILITY:
Inclusion Criteria:

* Minimum standards of physical activity proposed by the ACSM
* Perform running activity at high intensities (HIT)

Exclusion Criteria:

* No cardiovascular problems, respiratory or metabolic
* No muscle or joint injuries
* Not to use drugs or ergogenic resources

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2Max) | 0 week - 3 week (2 sessions for week)
  VO2Max measured in baseline and after training

SECONDARY OUTCOMES:
Time to Exhaustion (TLim 1% and 10%) | 0 week - 3 week (2 sessions for week)
  TLim1% and TLim10% Metabolically balanced (ACSM equation) measured in baseline and after training
Transfer of performance gains of TLim1% and TLim10% slope | 0 week - 3 week (2 sessions for week)
  Transfer of performance gains in TLim 1% and 10% slope
Peak Velocity | 0 week - 3 week (2 sessions for week)
  Performance in Progressive Test

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Machado, PhD, Study Director — Universidade Federal do Rio de Janeiro